CLINICAL TRIAL: NCT03564405
Title: A Open, Single-arm, Uncontrolled, Single Center, Pilot Study to Evaluate the Efficacy and Safety of UNI-DEB for Unresectable Hepatocellular Carcinoma
Brief Title: Pilot Clinical Trial to Evaluate the UNI-DEB for Unresectable Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNI-DEB-Pilot
Record Dates: First submitted 2018-06-11; First posted 2018-06-20 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Hepatocellular Carcinoma Non-resectable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UNI-DEB (Experimental)
  Interventions: Device: UNI-DEB

INTERVENTIONS:
Device: UNI-DEB — Applicate the TACE with UNI-DEB to unresectable hepatocellular carcinoma patient

SUMMARY:
Pilot Clinical Trial to Evaluate the Efficacy and Safety of UNI-DEB for Unresectable Hepatocellular Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Over 19 years
* Diagnosis of HCC
* Unresectable asymtomatic uninodular or multinodular tumor.
* Subject who maintain clinically normal hepatopetal flow without main portal vein closure
* At least one measurable target lesion by CT or MRI which 10 mm or more.
* ECOG Performance Status of 0 or 1.
* Child-Pugh class A or B
* Life expectancy of at least 6 months.

Exclusion Criteria:

* Another primary tumour, with the exception of conventional basal cell carcinoma or superficial bladder neoplasia
* Hepatic resection, liver transplantation or Percutaneous local treatment
* Previously received HCC related medical procedure
* Previously treated with anthracyclines
* Only measurable disease is within an area of the liver previously subjected to radiotherapy.
* Child Pugh C
* Active gastrointestinal bleeding within 6 months from screening.
* Total bilirubin > 3mg/dL
* WBC < 3,000cells/mm3
* ANC < 1,500cells/mm3
* Platelet < 50,000mm3
* Serum creatinine > 2mg/dL
* INR > 1.4
* ALT and AST > 5 times UNL
* Diffuse HCC defined as >50% tumor involvement of the whole liver.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 4 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University Seoul St. Mary Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No